CLINICAL TRIAL: NCT06982989
Title: Clinical Study on the Treatment of Pelvic Pain With Wearable Dual-band LED Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LED Pelvic pain; 2022YFB3604705 (Other Grant/Funding Number: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Pain
Keywords: LED; pelvic pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use LED to treat pelvic pain (Other): patient choose LED to treat pelvic pain
  Interventions: Device: use LED to treat pelvic pain

INTERVENTIONS:
Device: use LED to treat pelvic pain — Use led to treat pelvic pain

SUMMARY:
This study is a prospective clinical trial, which intends to prospective include female pelvic pain (dysmenorrhea and chronic pelvic pain), screen suitable cases, wear dual-band LED devices in non-menstrual period, perform low-dose phototherapy on local pelvic area and acupoints, and observe the changes of pelvic pain and related serological indicators in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* pelvic pain

Exclusion Criteria:

* Irregular menstrual cycles;
* Inflammatory disease;
* pregnant;
* Light allergy;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy that LED release pelvic pain | 1 month after the treatment
  Use VAS scale to evaluate the pain.The changes in the VAS score of pelvic pain before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Unniversity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT06982989/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT06982989/ICF_001.pdf